CLINICAL TRIAL: NCT04823403
Title: A Phase I Study Evaluating Safety and Efficacy of Hepatic Intra-Arterial Administration of Ipilimumab in Combination With Intra-venous Nivolumab for Advanced Hepatocellular Carcinoma
Brief Title: Hepatic Intra-Arterial Administration of Ipilimumab in Combination With Intra-venous Nivolumab for Advanced Hepatocellular Carcinoma
Acronym: HIPANIV
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-003766-40; 2020/3138 (Other: CSET number)
Record Dates: First submitted 2021-03-29; First posted 2021-03-30 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: Phase 1, Dose-Escalation (3+3 design), Open-label, single arm, single-center study, and expansion cohort. DLT will be captured within 1 month after HIA administration.
  3 levels of dose of HIA ipilimumab will be tested. Starting by a dose 5 times lower than what is used for IV administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with hepatocellular carcinoma (Experimental): 1. Intravenous Nivolumab (1mg/kg) will be given every 6 weeks for a maximal period of 6 months within the study.
  2. Ipilimumab, single intra-arterial (IA) injection per patient, at 3 dose-levels*.
     * (D1) Starting dose : 50 mg; n=3 to 6
     * (D2) 2nd dose-level : 100 mg; n=3 to 6
     * (D3) Maximal tested dose : 150mg; n=3 to 6 (if no limiting toxicities) *Dose level (D-1) : 25 mg will be tested if de-escalation is needed at D1 (>1/3 DLT at D1)
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Intravenous Nivolumab (1mg/kg) will be given every 6 weeks for a maximal period of 6 months within the study.
Drug: Ipilimumab — Ipilimumab, single intra-arterial (IA) injection per patient, at 3 dose-levels*.
  * (D1) Starting dose : 50 mg; n=3 to 6
  * (D2) 2nd dose-level : 100 mg; n=3 to 6
  * (D3) Maximal tested dose : 150mg; n=3 to 6 (if no limiting toxicities) *Dose level (D-1) : 25 mg will be tested if de-escalation is needed at D1 (>1/3 DLT at D1)

SUMMARY:
To determine the Maximum Tolerated Dose (MTD), and the recommended Phase 2 dose of HIA Ipilimumab in combination with IV Nivolumab by monitoring the Dose Limiting Toxicity (DLT) within 1 month after IA Ipilimumab administration in dose-escalation phase.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Men and women ≥ 18 years old
2. Patient should understand, sign, and date the written informed consent form prior to any protocol-specific procedures performed.
3. Patient should be able to comply with treatment, PK, and pharmacodynamic sample collection and willing to comply with study visits and procedures as per protocol.
4. Patients must have pathological confirmation of HCC.
5. Patient should be considered as non resectable by Multidisciplinary Team and liver surgeon, and non-eligible for liver transplantation (advanced HCC, BCLC C).
6. Patient who progresses on, or is intolerant to, or has refused standard first line therapy and eligible for receiving IV infusion of Nivolumab and HIA administration of Ipilimumab
7. Patient with active intrahepatic HCC. Part of the disease should not have undergone local treatments (including chemoembolization, or percutaneous targeted therapies).
8. Patients with or without active viral infection (i.e., HCV, HBV) are eligible. Patients with active HBV/HCV are eligible provided they are adequately treated to control the disease.
9. Patients should have measurable disease as defined by mRECIST criteria for response assessment.
10. ECOG status of 0 or 1 (Appendix 2).
11. Life expectancy of ≥ 12 weeks at the time of informed consent per Investigator assessment.
12. Adequate organ function as defined by the following:

    1. White blood cells (WBCs) ≥ 2000/mL
    2. Neutrophils ≥ 1000/mL
    3. Platelets ≥ 75 × 103/mL
    4. Hemoglobin ≥ 8.0 g/dL
    5. Creatinine < 1.5 × ULN or creatinine clearance ≥ 40mL/min (Cockcroft-Gault formula)
    6. ALT and AST ≤ 3 × ULN or < 5 x ULN in case of liver metastasis
    7. Lipase and amylase ≤ 1.5 × ULN
    8. Total bilirubin ≤ 1.5 × ULN
    9. Normal thyroid function, or stable on hormone supplementation per investigator assessment
13. Child-Pugh A, Without history of encephalopathy or clinically significant ascites
14. Women of childbearing potential (WOCBP) must have a negative urine or serum β-HCG pregnancy test within 14 days prior inclusion. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Sexually active female patients must agree to use two methods of effective contraception, one of them being a barrier method, or to abstain from sexual activity during the study and for at least 5 months after last study drug administration or must refrain from heterosexual activity during this same period.
15. Sexually active males patients must agree to use condom during the study and for at least 7 months after the last study treatment administration. Also, it is recommended their women of childbearing potential partner use a highly effective method of contraception for the same duration.
16. Patients shall be eligible to undergo pre-treatment and on-treatment tumor biopsies. Patients who either do not consent to a pre-treatment tumor biopsy or do not have accessible lesions will not be eligible.
17. Resolved acute effects of any prior therapy to baseline severity or NCI CTCAE v5 Grade ≤1 except for AEs not constituting a safety risk by investigator judgment.
18. Patients must be affiliated to a social security system or beneficiary of the same

Exclusion Criteria:

1. Patients with a prior malignancy are excluded, except those with prior malignancies treated more than 2 years previously (at the time of informed consent) with curative intent with no evidence of disease during the interval and who are considered by the Investigator to present a low risk for recurrence, will be eligible.
2. Patients with any active autoimmune disease or history of known or suspected autoimmune disease with the exception of patients with vitiligo, resolved/controlled asthma/atopy, controlled hypoadrenalism or hypopituitarism, and euthyroid patients with a history of Grave-Basedow"s disease (patients with controlled hyperthyroidism must be negative for thyroglobulin and thyroid peroxidase antibodies and thyroid stimulating immunoglobulin prior to inclusion).
3. A known or underlying medical condition that, in the opinion of the Investigator, could make the administration of study drug hazardous to the subject or could adversely affect the ability of the subject to comply with or tolerate study.
4. Requirement for daily supplemental oxygen
5. Any of the following within the 6 months prior to study entry: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack.
6. A confirmed history of encephalitis, meningitis, or uncontrolled seizures in the year prior to informed consent.
7. Positive blood screen for human immunodeficiency virus (HIV) with acquired immunodeficiency syndrome (AIDS). Patients with controlled HIV infection under anti-retroviral therapy and normal CD4+ T-cell counts (>500/mm3) could be considered eligible by the investigator if the patient fulfills the other inclusion/exclusion criteria.
8. Evidence of active infection that requires systemic antibacterial, antiviral, or antifungal therapy ≤ 7 days prior to inclusion.
9. Any other significant acute or chronic medical illness. Any other sound medical, psychiatric, and/or social reason as determined by the Investigator.
10. Subjects who are unable to undergo and/or tolerate venous AND arterial access (evaluated on pre-treatment imaging)
11. Systemic or topical corticosteroids at immunosuppressive doses (≥ 10 mg/day of prednisone or equivalent)
12. Patients that have received within 4 weeks or 5 half-lives (whichever is shorter) from inclusion and who are planned to receive the following during treatment:

    1. Any other investigational drug
    2. Any anticancer therapy (chemotherapy, biologics, therapeutic vaccines, radiotherapy, or hormonal treatment).
    3. Vaccines containing live virus
    4. Allergen hyposensitization therapy
    5. Growth factors, e.g., granulocyte-colony stimulating factor (G-CSF), granulocyte macrophage-colony stimulating factor (GM-CSF), erythropoietin
    6. Major surgery
    7. Bisphosphonates or anti-RANKL therapy
13. Previous allogeneic hematopoietic stem cell transplantation or previous solid organ transplantation requiring systemic immunosuppressive therapy
14. History of severe allergy, anaphylactic or other hypersensitivity reactions to chimeric or humanized antibodies or to biopharmaceutical produced in Chinese hamster ovarian cells or to any components of the study drugs
15. Patients with an active pneumonitis or a history of grade 3 or 4 pneumonitis due to the administration of immunotherapies.
16. Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent
17. Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2020-11-13 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 28 days
  To determine the Maximum Tolerated Dose (MTD), and the recommended Phase 2 dose of HIA Ipilimumab in combination with IV Nivolumab by monitoring the Dose Limiting Toxicity (DLT) within 1 month after IA Ipilimumab administration in dose-escalation phase.

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, France